CLINICAL TRIAL: NCT02026479
Title: Glucocorticoid Postauricular Injection Treatment for Sudden Hearing Loss: a Multi-center, Opened, Randomized, Controlled Clinical Trial
Brief Title: Sudden Hearing Loss Multi-center Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Sheng Yu, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCRP201307
Record Dates: First submitted 2013-12-29; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Full-frequency Sudden Hearing Loss
Keywords: full-frequency sudden hearing loss; post auricular injection; glucocorticoid; multi-center
MeSH Terms: interventions — dexamethasone 21-phosphate; ginaton

ARMS (3):
- regular treatment comparator (Experimental): Ginaton
  Interventions: Drug: Ginaton
- Dexamethasone Phosphate low dose (Experimental): 5mg
  Interventions: Drug: Dexamethasone Phosphate
- Dexamethasone Phosphate high dose (Experimental): 10mg
  Interventions: Drug: Dexamethasone Phosphate

INTERVENTIONS:
Drug: Dexamethasone Phosphate — 5mg; postauricular injection
  Arms: Dexamethasone Phosphate low dose
Drug: Dexamethasone Phosphate — 10mg; postauricular injection
  Arms: Dexamethasone Phosphate high dose
Drug: Ginaton — 40mg/pill, 3times/day,oral
  Arms: regular treatment comparator

SUMMARY:
The incidence of sudden hearing loss is rising obviously resent year, Glucocorticoids have obtained obvious effect in the treatment of sudden deafness. Postauricular hypodermic injection is the latest findings in clinical work and a new noninvasive way of administration which is gradually expanding research. The aim of this experiment is to verify and explore the efficacy and safety of the postauricular injection treatment with different doses of Glucocorticoids.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years, less than 60 years old;
* patient with unilateral or bilateral（occured successively) acute sensorineural hearing loss(ASNHL) with onset 72hours or less ago. Mean hearing loss compared with the unaffected contralateral ear of at leat 60 dB;
* Primary presentation within 2weeks; standard treatment for 2 weeks;
* After 2weeks of standard treatment, sensorineural hearing loss (SHL) curative effect evaluation damaged frequencies >/=30 dB better than before;
* Written informed consent before participation in the study.

Exclusion Criteria:

SYSTEMIC DISEASE

* History of tuberculosis or positive purified protein derivative (PPD);
* Insulin-dependent diabetes mellitus;
* Hypertension, poor control of BP(SBP/DBP)>=140mmHg);
* History of rheumatic disease, e.g. rheumatoid arthritis, scleroderma, lupus, etc;
* Serious psychiatric disease or psychiatric reaction to corticosteroids;
* History of heart disease or transient ischemic attacks(TIAs);
* Prior treatment with chemotherapeutic or immunosuppressive drugs;
* Pancreatitis;
* Active peptic ulcer disease or history of gastrointestinal bleeding;
* History of HIV, Hepatitis B or C;
* Chronic kidney failure;
* Alcohol abuse;
* Active shingles;
* Severe osteoporosis or non-surgical aseptic necrosis of the hip;
* Without contraindication with glucocorticoid, ginaton, Batroxobin.

OTOLOGIC DISEASE

* History of Meniere's disease;
* History of chronic ear infection;
* Prior history of sudden sensorineural hearing loss (SSNHL);
* History of fluctuating hearing loss.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pure tone audiometry test | Days 30
  Average change in hearing loss in decibel(dB) between the baseline and D 30 for the three contiguous frequencies with the worst hearing loss, and the treatment efficiency of the 30th day.

SECONDARY OUTCOMES:
Tinnitus with Evaluation questionnaire | days 14,30,90
  Average change in hearing loss in dB between the baseline and D 14, 90 for the three contiguous frequencies with the worst hearing loss; the treatment efficiency of the D 14,90; the treatment efficiency of the tinnitus in D14, 30, 90.
Vertigo with Evaluation questionnaire | Day 14,30,90
  Average change in hearing loss in dB between the baseline and D 14, 90 for the three contiguous frequencies with the worst hearing loss; the treatment efficiency of the D 14,90; the treatment efficiency of the vertigo in D14, 30, 90.

OTHER OUTCOMES:
the records of adverse reaction and event | Day 2,4,7,14,30,90
  the rate of adverse reaction and event